CLINICAL TRIAL: NCT05065203
Title: Evaluation of Inpatient Sleep and Activity Following Childbirth
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, PSultan, Associate Professor, Stanford University
Other Study IDs: 60762
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Sleep
Keywords: Postpartum sleep

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postpartum patients: Women booked and have delivery of their child(ren) at Lucile Packard Children's Hospital
  Interventions: Procedure: planned or unplanned Cesarean, operative, or non operative delivery

INTERVENTIONS:
Procedure: planned or unplanned Cesarean, operative, or non operative delivery — All types of delivery

SUMMARY:
Sleep is critical to mental and physical health following childbirth. However, patients who are hospitalized for labor and delivery may be admitted for days with significant impacts on sleep levels. Little is known about sleep and activity levels in inpatients during nighttime and daytime following childbirth and how this may affect their mental and physical health and wellbeing. If abnormalities are identified, targeted interventions may be possible to optimize recovery following delivery.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* live pregnancy
* Single or multiple gestation
* all gestational ages

Exclusion Criteria:

* Weekend delivery
* admitted to critical care
* unable to speak or understand English
* known sleeping disorder
* opioid requirement prior to admission
* long term steroids use
* significant autoimmune or neurological disease
* significant psychiatric or neurodevelopment disorder

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All pregnant women booked to deliver their child(ren) at Lucile Packard Children's Hospital. Eligible and consenting patients enrolled will wear an Actigraph watch during their inpatient stay (from preoperative period if undergoing cesarean delivery or during labor if undergoing a planned vaginal delivery).
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Assessment of inpatient postpartum sleep using actigraphy | During inpatient stay (up to 7 days)
  Participants will wear an acitgraphy watch during their inpatient stay to measure sleep.

SECONDARY OUTCOMES:
Association between actigraphy data with inpatient and outpatient postpartum Patient Reported Outcome Measures (PROMs) | Day 1-7, 6 and 12 weeks
  Measurement of postpartum actigraphy data to associate with patient reported outcome measures (PROM) (ObsQoR-10, Edinburgh Postpartum Depression Score, WHO-QOL-BREF and Bergen Insomnia Scale Score) given by face to face then remote interview
Association between inpatient actigraphy data and patient demographic, medical, obstetric, psychiatric, neonatal and anesthetic factors | During inpatient stay and outpatient follow up (up to 7 days)
  Participants will wear an acitgraphy watch during their inpatient stay to measure physical activity and sleep.
Association between outpatient sleep data with patient demographic, medical, obstetric, psychiatric, neonatal and anesthetic factors | 6 and 12 weeks
  Participants will be interviewed at 6 and 12 weeks with PROM questions and sleep diaries to assess for association with demographic, medical obstetric, psychiatric neonatal and anaesthetic factors.
Association between objective (artigraphy) and subjective sleep assessment using diaries and PROMs | Day 1-7, 6 and 12 weeks
  Participants will wear an acitgraphy watch during their inpatient stay to measure physical activity and sleep. PROM survey data during inpatient day 1-7 and outpatient 6- 12 week interview.
Determine population norms of objective and subjective sleep measures in the postpartum population. | Day 1-7, 6 and 12 weeks
  Participants will wear an acitgraphy watch during their inpatient stay to measure physical activity and sleep. PROM survey data during inpatient day 1-7 and outpatient 6 and 12 week interview.
Association between inpatient sleep and physical activity, PROMs and peripartum course with longer term outpatient sleep measures | Day 1-7, 6 and 12 weeks
  Participants will wear an acitgraphy watch during their inpatient stay to measure physical activity and sleep. PROM survey data during inpatient day 1-7 and outpatient 6 and 12 week interview.

CONTACTS AND LOCATIONS:
Overall Officials: Pervez Sultan, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
The data collected from the watches will not be available to share with other researchers.
  Anonymous and aggregated data will be available for verification only on request.